CLINICAL TRIAL: NCT05704114
Title: A Prospective, Single-center, Pilot Study to Evaluate the Efficacy, Safety, and Tolerability of Tazarotene 0.045% Lotion (Arazlo) for Treating Postinflammatory Erythema and Postinflammatory Hyperpigmentation in Subjects With Acne
Brief Title: Tazarotene 0.045% Lotion for Treating PIE and PIH in Subjects With Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Emmy Graber (Other)
Responsible Party: Sponsor-Investigator, Dr. Emmy Graber, President of The Dermatology Institute of Boston, Principal Investigator, The Dermatology Institute of Boston
Organization: The Dermatology Institute of Boston (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIB-0201
Record Dates: First submitted 2021-02-05; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Acne Vulgaris; Post Inflammatory Hyperpigmentation; Post Inflammatory Pigmentation Change; Erythema; Skin Scarring
Keywords: Acne vulgaris; Post Inflammatory Hyperpigmentation; Post Inflammatory Pigmentation Change; Erythema; Acne scars
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation; Erythema; Cicatrix | interventions — tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): This is a single arm study. All participants are receiving the treatment.
  Interventions: Drug: Tazarotene 0.045% Lotion

INTERVENTIONS:
Drug: Tazarotene 0.045% Lotion — Daily topical use of tazarotene for 16 weeks.
  Other Names: Arazlo

SUMMARY:
The purpose of the study is to assess the safety and efficacy of Arazlo Lotion (Tazarotene 0.045% Lotion) for treatment of postinflammatory erythema and postinflammatory hyperpigmentation in subjects with acne.

DETAILED DESCRIPTION:
This research study is studying Arazlo Lotion (Tazarotene 0.045% Lotion) as a possible treatment for treating postinflammatory erythema (skin reddening) and postinflammatory hyperpigmentation (dark skin spots) secondary to acne. Up to 20 people at the study doctor's office will be enrolled. Bausch Health USA is manufacturing the study drug in this research study.

The participants are being asked to participate in this research study because the participants have postinflammatory erythema and/or postinflammatory hyperpigmentation secondary to acne.

Postinflammatory erythema (PIE) is defined as the blanchable (turns white when pressed) red or pink macule (discolored spot) seen after an acne lesion (skin sore) resolves. PIE has been considered to be stage I scarring by some; however, PIE is not permanent but may be the preceding lesion for some atrophic (indented) scars. PIE is exceedingly common and is seen more in lighter skin types (I-III) and is often incorrectly considered by health care providers to be hyperpigmentation. PIE is nearly ubiquitous in acne patients with fairer skin tones and is blanchable erythema rather than hyperpigmentation. It differs from postinflammatory hyperpigmentation (PIH), which is the formation of dark macules due to an overexpression of melanin (dark pigment) that is secondary to an inflammatory response. PIH is particularly common in dark-skinned individuals.

PIE has been reportedly treated with in office treatments such as: pulsed dye laser, 1,450-nm laser, or fractional microneedling with radiofrequency; however, these treatments are not perfect. They come at a high financial cost to the patient, are not without side effects, are not well studied, and their efficacy for PIE is questionable. There is no known topical treatment for PIE that is secondary to acne. Conversely, various topicals do exist to treat PIH that work by inhibiting tyrosinase (an enzyme responsible for the first step in producing melanin), such as topical retinoids (compounds similar to Vitamin A). One small study showed tazarotene 0.1% cream to be effective in improving PIH. However, there are also reports of tazarotene worsening PIH, likely due to the skin irritation caused by the high strength of the tazarotene.

Our intended purpose is to demonstrate that Arazlo Lotion can reduce the formation of PIE and PIH in acne patients. The investigators hypothesize that Arazlo Lotion prevents the formation of PIE and PIH and treats PIE and PIH from acne due to its anti-inflammatory properties. These same anti-inflammatory properties of topical retinoids have been proven to reduce active acne lesions. However, no one has investigated the role of Arazlo Lotion on PIE and PIH. Small studies have shown that tazarotene 0.1% have improved PIH but other case reports have shown it to cause PIH. Utilizing Arazlo Lotion, a lower strength of tazarotene, in a gentler formulation, the investigators believe will lessen PIH without causing irritation and therefore reduce any potential PIH sequelae (conditions).

A participant cannot join this study if the participant has more than 3 excoriated (picked lesions) acne lesions, a beard or extensive facial hair, are a female subject who is pregnant, nursing, or planning a pregnancy during the trial, or the study doctor feels the participant needs to be treated with acne medications that are taken by mouth (also called "oral" medications). This is a study for subjects with discoloration, PIE and PIH, secondary to acne. The goal of treatment in this study is for the participant's acne discoloration to improve, which is no different than if the participant were to see the study doctor without being in the study.

The participant will receive the study drug, Arazlo Lotion, and any other topicals (applied on the skin) required by the study and all study examinations at no charge. The participant will receive payment to cover the costs of the participant's time and expenses to go to the study doctor's office for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, 18-45 years of age inclusive at Screening.
* Must have a facial IGA score of 2,3, or 4.
* Minimum of 10 inflammatory lesions (papules, pustules, or nodules) in total on face (including nose).
* Minimum of 20 PIE or PIH macules in total on face (including nose).
* Skin phototype of I to VI on Fitzpatrick's scale.
* Female subjects of childbearing potential must be on one of the following forms of birth control: a hormonal or non-hormonal IUD, an oral contraceptive pill that contains both estrogen and progestin, a contraceptive implant, or Depo shot. Patients will remain on the same contraception for 90 days prior to the baseline visit, for the duration of the study and for 1 month after.

Exclusion Criteria:

* More than 3 excoriated acne lesions.
* Beard or extensive facial hair.
* Female subject who is pregnant, nursing, or planning a pregnancy during the trial or within one month after last trial treatment application.
* Isotretinoin within 90 days.
* Other topical prescription retinoids (30 days wash out).
* A new hormone or hormone regulating therapy (such as spironolactone or birth control), or change in an existing dosage, for any reason within 90 days prior to screening. A patient who has been using the same regimen for more than 90 days prior to the study may be enrolled but is expected to remain on said regimen for the duration of the study.
* A new oral antibiotic or change in an existing dosage for any reason within 30 days prior to screening. A patient who has been using the same regiment for more than 30 days prior to the study may be enrolled but is expected to remain on the said regimen for the duration of the study.
* A new or change in topical anti-acne agents within 60 days of starting the study. This includes topical medications such as: benzoyl peroxide, erythromycin, clindamycin, minocycline, clascoterone, and dapsone. Use of such agents is permitted as long as subjects have been using these topical agents for at least 60 days prior and willing to stay on them for the duration of the study.
* Sebacia laser treatment within 180 days of study enrollment. Subjects may not have this treatment during the study.
* Any facial laser treatment or chemical peel within one month of enrollment. Subjects may not have these treatments during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Reduction of postinflammatory erythema lesion count. | 16 weeks
  A count of postinflammatory erythema lesions will be conducted at each visit.
Reduction of postinflammatory hyperpigmentation lesion count. | 16 weeks
  A count of postinflammatory hyperpigmentation lesions will be conducted at each visit.
Reduction of active acne lesion count | 16 weeks
  Active acne lesions will be counted at each visit.

SECONDARY OUTCOMES:
Patient perceived improvement through completion of a patient satisfaction survey | 16 weeks
  The patient will fill out a questionnaire at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Emmy Graber, Principal Investigator — The Dermatology Insitutue of Boston
Locations (1):
- The Dermatology Institute of Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Tan J, Bourdes V, Bissonnette R, Petit B Eng L, Reynier P, Khammari A, Dreno B. Prospective Study of Pathogenesis of Atrophic Acne Scars and Role of Macular Erythema. J Drugs Dermatol. 2017 Jun 1;16(6):566-572. PMID 28686774
- [Result] Fabbrocini G, Annunziata MC, D'Arco V, De Vita V, Lodi G, Mauriello MC, Pastore F, Monfrecola G. Acne scars: pathogenesis, classification and treatment. Dermatol Res Pract. 2010;2010:893080. doi: 10.1155/2010/893080. Epub 2010 Oct 14. PMID 20981308